CLINICAL TRIAL: NCT00595738
Title: Use of Peripheral Venous Oxygen Saturation and Biomarkers to Estimate Cardiac Output and Filling Pressures in Patients With Advanced Heart Failure
Brief Title: Peripheral Venous Oxygen Saturation and Biomarkers to Estimate Cardiac Output and Filling Pressures in Heart Failure
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Siemens Molecular Imaging (Industry); Critical Diagnostics (Industry)
Responsible Party: Thomas J. Wang, MD, Massachusetts General Hospital
Other Study IDs: 2007P-000704
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Congestive Heart Failure
Keywords: Congestive heart failure; Cardiac biomarkers; Hemodynamics; Tailored therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will be banking serum collected from peripheral blood draws, and blood draws from a pulmonary artery catheter and arterial line.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure Patients: Patients admitted with advanced heart failure for tailoring of heart failure therapy via placement of a pulmonary artery (PA) catheter. In our study, the patients will already have a PA catheter placed for clinical/treatment reasons when we approach them for the study.
  Interventions: Other: Standard of care therapy for severe decompensated heart failure

INTERVENTIONS:
Other: Standard of care therapy for severe decompensated heart failure — Standard of care therapy for severe decompensated heart failure

SUMMARY:
The relationship between peripheral venous saturation and central hemodynamics (including right and left heart filling pressures and cardiac output), mixed venous oxygen saturation, and contemporary biomarkers of heart failure is not clear. We aim to determine the relationship between mixed venous, central venous, and peripheral venous oxygen saturation in patients with advanced (class III or IV) heart failure. We will determine the relationship between cardiac output measured via thermodilution and the Fick equation calculated using concurrent oxygen saturations from the distal PA, central vein, and peripheral vein. We also aim to examine the relationship of selected cardiac biomarkers with cardiac filling pressures and cardiac output over time in patients with decompensated heart failure.

ELIGIBILITY:
The following inclusion criteria will be utilized:

1. Age>21
2. PA-catheter insertion for therapy of congestive heart failure decided upon by the attending cardiologist

The following will be considered as exclusion criteria for this study

1. Known or suspected septic shock or bacteremia
2. Active bleeding or HCT<24% at baseline
3. Arterial oxygen saturation <90% at baseline despite supplemental oxygen therapy.
4. Previous difficulty with venipuncture of upper extremity veins or the presence of a surgical arteriovenous fistula for hemodialysis
5. Insertion of the PA catheter through the femoral vein
6. Subjects unwilling or unable to provide written consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 30 patients admitted to the Massachusetts General Hospital Coronary Care Unit (CCU) for PA catheter-directed therapy for advanced heart failure. Only patients for whom the attending cardiologist has already decided upon PA-catheter insertion will be recruited for the study.
  Potential subjects will be identified by the CCU attending cardiologist, and a study nurse will review each patient for the exclusion criteria as above. Final decisions on patient eligibility will be made by Dr. Wang.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the relationship between mixed venous, central venous, and peripheral venous oxygen saturation in patients with advanced (class III or IV) heart failure. | Day 0-5 of 'tailored' heart failure therapy

SECONDARY OUTCOMES:
To examine the relationship of selected cardiac biomarkers with cardiac filling pressures and cardiac output over time in patients with decompensated heart failure. | Days 0-5 of 'tailored' heart failure therapy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Wang, MD, Principal Investigator — Massachusetts General Hospital; James Januzzi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Coronary Care Unit, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zilinski JL, Shah RV, Gaggin HK, Gantzer ML, Wang TJ, Januzzi JL. Measurement of multiple biomarkers in advanced stage heart failure patients treated with pulmonary artery catheter guided therapy. Crit Care. 2012 Jul 25;16(4):R135. doi: 10.1186/cc11440. PMID 22830581